CLINICAL TRIAL: NCT00101608
Title: A Phase II Study of Intravenous (IV) Vinflunine in Patients With Locally Advanced or Metastatic Transitional Cell Carcinoma (TCC) of the Urothelium
Brief Title: Vinflunine in Patients With Locally Advanced or Metastatic Transitional Cell Carcinoma of the Urothelium
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Pierre Fabre Medicament (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA183-001; NCT00268424 (obsolete NCT alias)
Record Dates: First submitted 2005-01-12; First posted 2005-01-13 (Estimated); Last update posted 2010-03-02 (Estimated); Status verified 2008-08

CONDITIONS: Transitional Cell Carcinoma; Bladder Neoplasms; Kidney Neoplasms; Ureter Neoplasms; Bladder Cancer; Neoplasm, Bladder
Keywords: urothelium
MeSH Terms: conditions — Carcinoma, Transitional Cell; Urinary Bladder Neoplasms; Kidney Neoplasms; Ureteral Neoplasms | interventions — vinflunine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: vinflunine

INTERVENTIONS:
Drug: vinflunine — solution for injection, IV, 280/320 mg/m2, every 3 wks, variable duration

SUMMARY:
The purpose of this clinical research study is to learn if vinflunine can shrink or slow the growth of the cancer or increase survival in patients with transitional cell carcinoma of the urothelium. The safety of this treatment will also be studied.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of transitional cell carcinoma of the urothelium that is locally advanced or metastatic (i.e. patients cannot be candidates for local/regional control of disease).
* Relapse or progression within 12.5 months of prior cisplatin or carboplatin containing chemotherapy regimen.
* Adequate performance status (Karnofsky greater or equal to 80).

Exclusion Criteria:

* Receipt of more than 1 prior chemotherapy regimen in any setting.
* Prior discontinuation of platinum due solely to toxicity.
* Current neuropathy greater or equal to CTC grade 2.
* Prior radiation to greater or equal to 30% of bone marrow.
* Inadequate hematologic function: ANC <1,500 cells/mm3, Platelet<100,000 cells/mm3.
* Inadequate hepatic function: total bilirubin > 1.5 times ULN, ALT/AST > 2.5 times ULN or > 5 times ULN in case of liver metastasis.
* Inadequate renal function: creatinine clearance <20 ml/min.
* Prior allergy to any vinca-alkaloid.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2005-01; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
To estimate the objective response rate in patients with TCC of the urothelium receiving vinflunine, who had evidence of documented progression at any time within 12 months after the last dose of platinum therapy and are not candidates of cystectomy. | 10-Apr-2007

SECONDARY OUTCOMES:
To estimate duration of response, time to response disease control rate, progression free survival, and overall survival in this patient population, and evaluate the safety profile of vinflunine | 10-April-2007

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (75):
- United States (38):
  - Local Institution, Beverly Hills, California
  - Local Institution, La Jolla, California
  - Local Institution, Los Angeles, California
  - Local Institution, Santa Monica, California
  - Local Institution, Stanford, California
  - Local Institution, Vallejo, California
  - Local Institution, Aurora, Colorado
  - Local Institution, New Haven, Connecticut
  - Local Institution, Washington D.C., District of Columbia
  - Local Institution, Jacksonville, Florida
  - Local Institution, Miami, Florida
  - Local Institution, Atlanta, Georgia
  - Local Institution, Honolulu, Hawaii
  - Local Institution, Chicago, Illinois
  - Local Institution, Joliet, Illinois
  - Local Institution, Urbana, Illinois
  - Local Institution, Louisville, Kentucky
  - Local Institution, Baltimore, Maryland
  - Local Institution, Burlington, Massachusetts
  - Local Institution, Ann Arbor, Michigan
  - Local Institution, Detroit, Michigan
  - Local Institution, Kansas City, Missouri
  - Local Institution, St Louis, Missouri
  - Local Institution, Las Vegas, Nevada
  - Local Institution, Lebanon, New Hampshire
  - Local Institution, Buffalo, New York
  - Local Institution, New York, New York
  - Local Institution, The Bronx, New York
  - Local Institution, Charlotte, North Carolina
  - Local Institution, Durham, North Carolina
  - Local Institution, Cincinnati, Ohio
  - Local Institution, Philadelphia, Pennsylvania
  - Local Institution, Pittsburgh, Pennsylvania
  - Local Institution, Providence, Rhode Island
  - Local Institution, Nashville, Tennessee
  - Local Institution, Dallas, Texas
  - Local Institution, Seattle, Washington
  - Local Institution, Milwaukee, Wisconsin
- Australia (6):
  - Local Institution, Liverpool, New South Wales
  - Local Institution, Sydney, New South Wales
  - Local Institution, Taree, New South Wales
  - Local Institution, Waratah, New South Wales
  - Local Institution, Westmead, New South Wales
  - Local Institution, Adelaide, South Australia
- Austria (2):
  - Local Institution, Linz
  - Local Institution, Salzburg
- Canada (4):
  - Local Institution, Edmonton, Alberta
  - Local Institution, London, Ontario
  - Local Insitution, Toronto, Ontario
  - Local Institution, Montreal, Quebec
- France (5):
  - Local Institution, Caen
  - Local Institution, Le Mans
  - Local Institution, Nice
  - Local Institution, Paris
  - Local Institution, Toulouse
- Local Institution, Nea Liosia, Greece
- Local Institution, Jakarta, Indonesia
- Italy (5):
  - Local Institution, Genova
  - Local Institution, Milan
  - Local Institution, Roma
  - Local Institution, Rome
  - Local Institution, Viterbo
- Philippines (3):
  - Local Institution, Cebu City
  - Local Institution, Quezon
  - Local Institution, Quezon City
- Local Institution, Singapore, Singapore
- Local Institution, Seoul, South Korea
- Spain (4):
  - Local Institution, Murcia
  - Local Institution, Palma de Mallorca
  - Local Institution, Santander
  - Local Institution, Seville
- Sweden (2):
  - Local Institution, Linköping
  - Local Institution, Uppsala
- Local Institution, Aarau, Switzerland
- Local Institution, Bangkok, Thailand